CLINICAL TRIAL: NCT01996306
Title: A Multinational, Randomized, Phase III Study of XELIRI With/Without Bevacizumab Versus FOLFIRI With/Without Bevacizumab As Second-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: A Phase III Study of 2nd-line XELIRI ± Bevacizumab vs. FOLFIRI ± Bevacizumab in mCRC
Acronym: AXEPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AXEPT; UMIN000012263 (Other: UMIN)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms
Keywords: AXEPT; Fluorouracil; CPT-11; XELIRI; Bevacizumab; FOLFIRI; Capecitabine; 2nd-line metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — Bevacizumab; Irinotecan; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRI +/- Bevacizumab (Active Comparator): Bevacizumab 5 mg/kg IV 90-30 min Day 1 CPT-11 180 mg/m2 (150 mg/m2) IV 90 min Day 1 l-LV (dl-LV) 200 mg/m2 (400 mg/m2) IV 120 min Day 1 5-FU - bolus 400 mg/m2 IV bolus Day 1 5-FU - infusional 2400 mg/m2 IV continuous (46 hours) Day 1 - 3
  Interventions: Biological: Bevacizumab; Drug: CPT-11 (Irinotecan); Drug: 5-FU Bolus; Drug: 5-FU Infusion; Drug: l-LV (dl-LV)
- XELIRI +/- Bevacizumab (Experimental): Bevacizumab 7.5 mg/kg IV 90-30 min Day 1 CPT-11 200 mg/m2 (150 mg/m2) IV 90 min Day 1 Capecitabine 800 mg/m2 p.o. twice daily 14 Days consecutively
  Interventions: Biological: bevacizumab; Drug: CPT-11 (Irinotecan); Drug: Capecitabine

INTERVENTIONS:
Biological: Bevacizumab — 5 mg/kg intravenously administered over 90 minutes (can be reduced to 30 minutes at the minimum) on day 1 of a 2-week cycle.
  Other Names: Avastin
  Arms: FOLFIRI +/- Bevacizumab
Drug: CPT-11 (Irinotecan) — 150-180 mg/m2 intravenously administered over 90 minutes on day 1 of a 2-week cycle.
  Other Names: Irinotecan
  Arms: FOLFIRI +/- Bevacizumab
Drug: 5-FU Bolus — 400 mg/m2 intravenous bolus on day 1 of a 2-week cycle.
  Other Names: fluorouracil
  Arms: FOLFIRI +/- Bevacizumab
Drug: 5-FU Infusion — 2400 mg/m2 continuous infusion over 46 hours on day 1 and 2 of a 2-week cycle.
  Other Names: fluorouracil
  Arms: FOLFIRI +/- Bevacizumab
Drug: l-LV (dl-LV) — 200 (dl-LV: 400) mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle.
  Other Names: Leucovorin
  Arms: FOLFIRI +/- Bevacizumab
Biological: bevacizumab — 7.5mg/kg IV intravenously administered over 90 minutes (can be reduced to 30 minutes at the minimum) on Day 1 of a 3-week cycle.
  Other Names: Avastin
  Arms: XELIRI +/- Bevacizumab
Drug: CPT-11 (Irinotecan) — 150-200 mg/m2 intravenously administered over 90 minutes on day 1 of a 3-week cycle.
  Other Names: Irinotecan
  Arms: XELIRI +/- Bevacizumab
Drug: Capecitabine — 1600mg/m2/day oral on day 1 (evening) to day 15 (morning)of a 3-week cycle.
  Other Names: Xeloda
  Arms: XELIRI +/- Bevacizumab

SUMMARY:
The primary purpose of this study is to determine the non-inferiority of overall survival XELIRI with or without Bevacizumab compared with FOLFIRI with or without Bevacizumab as Second-line therapy in Patient with Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
Primary endpoint: Overall survival (OS), Secondary endpoints: Progression-free survival (PFS), Time to treatment failure (TTF), Overall response rate (ORR),Disease Control Rate (DCR), Relative dose intensity, Safety, and Correlation between UGT1A1 genotype and Safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed inoperable colorectal adenocarcinoma excluding vermiform appendix cancer and anal canal cancer.
2. Age ≥20 years at the time of informed consent
3. ECOG performance status (PS) of 0-2
4. Written informed consent prior to study-specific screening procedures
5. Life expectancy of at least 90 days
6. Withdrawal from first-line chemotherapy (regardless of containing molecular-targeted drugs) for metastatic colorectal cancer due to intolerable toxicity or progressive disease, or relapse within 180 days after the last dose of adjuvant chemotherapy.
7. Adequate organ function according to following laboratory values obtained within 14 days before enrolment (excluding patients who received blood transfusions or hematopoietic growth factors within 14 days before the laboratory test) Neutrophil count: ≥1500/mm3 Platelet count: ≥10.0 x 104/mm3 Hemoglobin: ≥9.0 g/dL Total bilirubin: ≤1.5 mg/dL AST, ALT: ≤100 IU/L (≤200 IU/I if liver metastases present) Serum creatinine: ≤1.5 mg/dL

Exclusion Criteria:

1. History of other malignancy with a disease-free interval <5 years (other than curatively treated cutaneous basal cell carcinoma, curatively treated carcinoma in situ of the cervix, and gastroenterological cancer confirmed to be cured by endoscopic mucosal resection)
2. With massive pleural effusion or ascites requiring intervention
3. Radiological evidence of brain tumor or brain metastases
4. Active infection including hepatitis
5. Any of the following complication:

   i) Gastrointestinal bleeding or gastrointestinal obstruction (including paralytic ileus) ii) Symptomatic heart disease (including unstable angina, myocardial infarction, and heart failure) iii) Interstitial pneumonia or pulmonary fibrosis iv) Uncontrolled diabetes mellitus v) Uncontrolled diarrhea (that interferes with daily activities despite adequate therapy)
6. Any of the following medical history:

   Myocardial infarction: History of one episode within one year before enrollment or two or more lifetime episodes i) Serious hypersensitivity to any of the study drugs ii) History of adverse reaction to fluoropyrimidines suggesting dihydropyrimidine dehydrogenase (DPD) deficiency
7. Previous treatment with irinotecan hydrochloride
8. Current treatment with atazanavir sulfate
9. Previous treatment with tegafur, gimeracil, and oteracil potassium within seven days before enrollment
10. Pregnant or lactating females, and males and females unwilling to use contraception
11. Requires continuous treatment with systemic steroids
12. Psychiatric disability that would preclude study compliance
13. Otherwise determined by the investigator to be unsuitable for participation in the study
14. Concurrent gastrointestinal perforation or history of gastrointestinal perforation with 1 year before enrollment
15. History of pulmonary hemorrhage/hemoptysis ≥ Grade 2 (defined as bright red blood of at least 2.5mL) within 1 month prior to enrollment.
16. History of laparotomy, thoracotomy, or intestinal resection within 28 days before enrollment
17. Unhealed wound (except suture wounds from implantation of a central venous port), gastrointestinal ulcer, or traumatic fracture
18. Current or recent (within 1 year) thromboembolism or cerebrovascular disease
19. Currently receiving or requires anticoagulation therapy (> 325 mg/day of aspirin)
20. Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR ≥1.5 within 14 days before enrollment)
21. Uncontrolled hypertension
22. Urine dipstick for proteinuria >+2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.
Time to treatment failure (TTF) | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to the earlier of the date of confirmed progression, death from any cause, or discontinuation of protocol treatment.
Overall Response Rate (ORR) | Assessed at 6, 12 week and thereafter every 8 weeks
  Proportion of eligible patients with measurable lesions with a best overall response of CR or PR assessed by the attending physician.
Disease Control Rate (DCR) | Assessed at 6, 12 week and thereafter every 8 weeks
  Proportion of best overall response of CR, PR, or SD assessed by the attending physician.
Relative Dose Intensity | Assessed until final dosing to the last patient
  will be calculated for each drug to evaluate treatment compliance in the all-treated population during the observation period.
Incidence of Adverse Events (Adverse Reactions) | Adverse events occurring within 30 days after treatment discontinuation will be followed until recovery
  The incidence of worst-grade adverse events (toxicities) on study as graded by NCI-CTCAE v 4.0 will be determined by treatment arm in all treated patients for the following events.
Correlation between UGT1A1 genotype and safety | Adverse events occurring within 30 days after treatment discontinuation will be followed until recovery
  The incidence of worst-grade adverse events on study as graded by NCI-CTCAE v 4.0 will be determined by treatment arm and UGT1A1 genotype in all treated patients with a known UGT1A1 genotype profile

CONTACTS AND LOCATIONS:
Overall Officials: Kei Muro, MD, Principal Investigator — Aichi Cancer Center Hospital, Japan; Tae Won Kim, MD, PhD, Principal Investigator — ASAN Medical center, South Korea; Young Suk Park, MD, PhD, Principal Investigator — Samsung Medical Center, South Korea; Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-Sen University Cancer Center, China
Locations (1):
- NPO Epidemiological and Clinical Research Information Network (ECRIN), Kyoto, Japan

REFERENCES:
- [Derived] Xu RH, Muro K, Morita S, Iwasa S, Han SW, Wang W, Kotaka M, Nakamura M, Ahn JB, Deng YH, Kato T, Cho SH, Ba Y, Matsuoka H, Lee KW, Zhang T, Yamada Y, Sakamoto J, Park YS, Kim TW. Modified XELIRI (capecitabine plus irinotecan) versus FOLFIRI (leucovorin, fluorouracil, and irinotecan), both either with or without bevacizumab, as second-line therapy for metastatic colorectal cancer (AXEPT): a multicentre, open-label, randomised, non-inferiority, phase 3 trial. Lancet Oncol. 2018 May;19(5):660-671. doi: 10.1016/S1470-2045(18)30140-2. Epub 2018 Mar 16. PMID 29555258
- [Derived] Kotaka M, Xu R, Muro K, Park YS, Morita S, Iwasa S, Uetake H, Nishina T, Nozawa H, Matsumoto H, Yamazaki K, Han SW, Wang W, Ahn JB, Deng Y, Cho SH, Ba Y, Lee KW, Zhang T, Satoh T, Buyse ME, Ryoo BY, Shen L, Sakamoto J, Kim TW. Study protocol of the Asian XELIRI ProjecT (AXEPT): a multinational, randomized, non-inferiority, phase III trial of second-line chemotherapy for metastatic colorectal cancer, comparing the efficacy and safety of XELIRI with or without bevacizumab versus FOLFIRI with or without bevacizumab. Chin J Cancer. 2016 Dec 22;35(1):102. doi: 10.1186/s40880-016-0166-3. PMID 28007025